CLINICAL TRIAL: NCT04655664
Title: The Use of the 25 (OH) D Saliva Test as a Substitute for the 25 (OH) D Serum Test in Healthy People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, DINA KEUMALA SARI, Principal Investigator, Universitas Sumatera Utara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: USumateraUtara 1
Record Dates: First submitted 2020-11-18; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Nutritional Deficiency
Keywords: vitamin D; cross-sectional; non-invasive; correlation; deficiency; insufficiency
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Men and women aged 18-60 years, not currently experiencing chronic pain, kidney problems, liver problems, or other hormone disorders
  Interventions: Diagnostic Test: not currently consumed vitamin D supplements regularly
- Regularly Group (Active Comparator): Subjects who consumed vitamin D supplements regularly, were pregnant, or were breastfeeding.
  Interventions: Diagnostic Test: consumed vitamin D supplements regularly

INTERVENTIONS:
Diagnostic Test: not currently consumed vitamin D supplements regularly — The tests carried out were examination of 25 (OH) D and 1.25 (OH) D levels of serum and saliva, examination of demographic data, and other anthropometries. The examination was carried out by taking 5 mL of blood and 2 mL of saliva, and then checking the serum and saliva levels of 25 (OH) D and 1.25 (OH) D. Before the examination, the research subjects were asked not to consume food or drink for at least 90 minutes before being examined. Centrifugation was carried out (2500 g, 10 minutes) and the product immediately stored at -20 oC. In the serum examination, after the blood was drawn, centrifugation was carried out and the product stored at -20 oC for further determination of the levels of 25 (OH) D and 1.25 (OH) saliva.
  Arms: Treatment Group
Diagnostic Test: consumed vitamin D supplements regularly — The tests carried out were examination of 25 (OH) D and 1.25 (OH) D levels of serum and saliva, examination of demographic data, and other anthropometries. The examination was carried out by taking 5 mL of blood and 2 mL of saliva, and then checking the serum and saliva levels of 25 (OH) D and 1.25 (OH) D. Before the examination, the research subjects were asked not to consume food or drink for at least 90 minutes before being examined. Centrifugation was carried out (2500 g, 10 minutes) and the product immediately stored at -20 oC. In the serum examination, after the blood was drawn, centrifugation was carried out and the product stored at -20 oC for further determination of the levels of 25 (OH) D and 1.25 (OH) saliva.
  Arms: Regularly Group

SUMMARY:
Routine examination of vitamin D levels is carried out by checking serum 25 (OH)D levels, which indicate circulating vitamin D levels. While serum 1.25 (OH) D levels are less frequently utilized, they represent the active form of vitamin D and could be a substitute for checking vitamin D levels. This study aims to find the correlation between vitamin D levels, namely 25 (OH) D and 1.25 (OH) D saliva, which correlate with serum 25 (OH) D and 1.25 (OH) D levels in the examination of salivary vitamin D, and which could be a substitute for checking serum vitamin D levels.

DETAILED DESCRIPTION:
Routine examination of vitamin D levels is carried out by checking serum 25 (OH)D levels, which indicate circulating vitamin D levels. While serum 1.25 (OH) D levels are less frequently utilized, they represent the active form of vitamin D and could be a substitute for checking vitamin D levels.This study aims to find the correlation between vitamin D levels, namely 25 (OH) D and 1.25 (OH) D saliva, which correlate with serum 25 (OH) D and 1.25 (OH) D levels in the examination of salivary vitamin D, and which could be a substitute for checking serum vitamin D levels.This study is a cross-sectional study involving healthy men and women, aged 20-50 years, from Lima Puluh Village, Batubara District, North Sumatra Province, Indonesia. The parameters studied were 25 (OH) D and 1.25 (OH) D levels of saliva and serum.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 18-60 years, not currently experiencing chronic pain, kidney problems, liver problems, or other hormone disorders.

Exclusion Criteria:

* subjects who consumed vitamin D supplements regularly, were pregnant, or were breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-04-11 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Salivary 25 (OH) D | up to 2 weeks
  Salivary 25 (OH) D assay can be used to replace serum 25 (OH) D assay in healthy people as a non-invasive alternative. Examination using saliva as a substitute for serum testing is expected to facilitate the examination of 25 (OH) D.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Universitas Sumatera Utara, Medan, North Sumatra, Indonesia

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT04655664/Prot_SAP_ICF_000.pdf